CLINICAL TRIAL: NCT02333669
Title: Association of SCNN1A Single Nucleotide Polymorphisms With Neonatal Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Li Wang, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: DapingH023
Record Dates: First submitted 2015-01-03; First posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Neonatal Respiratory Distress Syndrome
Keywords: Lung fluid absorption disorders; Neonatal respiratory distress syndrome; Single nucleotide polymorphism; SCNN1A
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control group: The control blood samples, which were collected from healthy neonatal umbilical cord blood, were obtained from the maternity ward of 80 hospitals in Chongqing and nearby areas
  Interventions: Other: no intervention
- RDS group: Newborns with RDS were consecutively recruited for this study from the neonatal intensive care unit (NICU) at Daping Hospital, Third Military Medical University, Chongqing, China, a tertiary care facility
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Lung fluid absorption disorders are largely mediated by transepithelial Na+ reabsorption through alpha epithelial sodium channels (α-ENaCs) in alveolar epithelial cells. Increasing evidence has demonstrated that these lung disorders might be an important cause of neonatal respiratory distress syndrome (NRDS) by influencing gas exchange or surfactant function, particularly in near-term and term infants. The SCNN1A gene, which encodes the α-ENaC, might predispose infants to NRDS. To explore whether the single-nucleotide polymorphisms (SNPs) of SCNN1A are associated with NRDS, we conducted a case-control study to investigate the NRDS-associated loci in Han Chinese infants. Seven target SNPs were selected from the SCNN1A gene and were genotyped using the improved multiplex ligase detection reaction (iMLDR).

ELIGIBILITY:
Inclusion Criteria:

* Newborns with RDS

Exclusion Criteria:

* The infants were excluded if they had any congenital malformation, inherited metabolic abnormalities, intrauterine infection, Rh/Rh incompatibility, pneumonia, pulmonary hypertension, meconium aspiration syndrome, or asphyxia

Ages: 1 Minute to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns with RDS are consecutively recruited for this study from the neonatal intensive care unit (NICU) at Daping Hospital, Third Military Medical University, Chongqing, China, a tertiary care facility. The control blood samples, which are collected from healthy neonatal umbilical cord blood, are obtained from the maternity ward of 80 hospitals in Chongqing and nearby areas.
Sampling Method: Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Genotype distributions of target SNPs in RDS group and Control group | within 28 days after birth
  Compare the genotype and allele frequencies of target SNPs between RDS group and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shi, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Department of pediatrics, Daping Hospital, The Third Military Medical University, Chongqing, Chongqing Municipality, China